CLINICAL TRIAL: NCT01857999
Title: Short-term add-on Therapy With Angiotensin Receptor Blocker for End-stage Inotrope-dependent Heart Failure Patients: B-type Natriuretic Peptide Reduction in a Randomized Clinical Trial
Brief Title: Losartan in Decompensated Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Marcelo Eidi Ochiai, Ph.D., InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCOR 2993/07/008
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2011-03

CONDITIONS: Congestive Heart Failure; Low Cardiac Output
Keywords: Renin-aldosterone system; Hemodynamic; Low cardiac output; Vasodilation; Natriuretic peptide
MeSH Terms: conditions — Heart Failure; Cardiac Output, Low; Aneurysm | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan (Experimental): Losartan 50 mg bid orally
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Placebo 1 pill bid orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan
  Arms: Losartan
Drug: Placebo
  Arms: Placebo

SUMMARY:
The dual blockade of the renin-angiotensin-aldosterone system with an angiotensin-converting enzyme inhibitor and an angiotensin-receptor blocker used together in heart failure patients has been demonstrated to be beneficial. However, the dual inhibition has not been studied during heart failure decompensation or even when low cardiac output is present.

The objective of this study was to assess the effects of add-on therapy with angiotensin receptor blocker on plasma B-type natriuretic peptide levels and hemodynamic measurements in heart failure patients with low cardiac output during hospitalization for decompensation.

This was a randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
The inclusion criteria were hospitalization for decompensated heart failure defined by worsening of symptoms until fatigue or dyspnea at rest, low cardiac output defined by the clinical-hemodynamic profile, dobutamine dependence, and ejection fraction < 0.45, spontaneous breathing and receiving angiotensin-converting enzyme inhibitors. The patients could have jugular ingurgitation, lower limbs edema, ascites and rales. Dobutamine dependence was defined by infusion for more than 15 days or an unsuccessful attempt of withdrawal.

The exclusion criteria were serum creatinine > 3.0 mg/dL, serum potassium > 6.0 mEq/L, systolic blood pressure < 70 mm Hg, aortic stenosis, and acute coronary syndrome in the previous 2 months. The patients were randomly assigned by permuted block of 4, stratified by sex, to losartan or placebo.

The endpoints were change in B-type natriuretic peptide levels, cardiac index, pulmonary wedge capillary pressure, systemic vascular resistance, and successful withdrawal of dobutamine.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization for decompensated heart failure
* dobutamine dependence
* ejection fraction < 0.45
* taking angiotensin-converting enzyme inhibitor

Exclusion Criteria:

* serum creatinine > 3.0 mg/dL
* serum potassium > 6.0 mEq/L
* systolic blood pressure < 70 mm Hg
* aortic stenosis
* acute coronary syndrome in the previous 2 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
B-type natriuretic peptide | 7 days
  Serum B-type natriuretic peptide

SECONDARY OUTCOMES:
Successful withdrawal from dobutamine | 7 days
  Successful withdrawal from dobutamine with clinical stability
Worsening renal function | 7 days
  Increase > 0.3 mg/dL in serum creatinine
Hyperkalemia | 7 days
  Serum potassium > 5.5 mEq/L
Hypotension | 7 days
  Systolic blood pressure < 80 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Antonio P Barretto, Ph.D., Study Director — Heart Institute (InCor), University of São Paulo
Locations (1):
- Cotoxó Hospital, Heart Institute (InCor), University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ochiai ME, Brancalhao EC, Puig RS, Vieira KR, Cardoso JN, Oliveira MT Jr, Barretto AC. Short-term add-on therapy with angiotensin receptor blocker for end-stage inotrope-dependent heart failure patients: B-type natriuretic peptide reduction in a randomized clinical trial. Clinics (Sao Paulo). 2014;69(5):308-13. doi: 10.6061/clinics/2014(05)02. PMID 24838894